CLINICAL TRIAL: NCT01523769
Title: The Efficacy of Umbilical Cord Milking on the Reduction of Red Blood Cell Transfusion Rates in Infants Born Between 24 and 28 6/7 Weeks Gestation, a Randomized Controlled Trial.
Brief Title: Umbilical Cord Milking on the Reduction of Red Blood Cell Transfusion Rates in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EasternVMC
Record Dates: First submitted 2011-12-16; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Prematurity
Keywords: prematurity; umbilical cord milking; delayed cord clamping; neonatal transfusion
MeSH Terms: conditions — Premature Birth | interventions — Umbilical Cord Clamping; Blood Transfusion, Autologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Control group, the cord was not milked
- Umbilical Cord Milking (Experimental): Approximately 10 cm of umbilical cord was milked toward the baby immediately following delivery
  Interventions: Procedure: Umbilical Cord Milking

INTERVENTIONS:
Procedure: Umbilical Cord Milking — Approximately 10 cm of umbilical cord was milked toward the baby immediately following delivery. (The blood remaining in the umbilical cord after delivery is squeezed in the direction from the placenta (remaining inside the uterus) toward the newborn baby.)
  Other Names: Umbilical Cord Milking, autotransfusion
  Arms: Umbilical Cord Milking

SUMMARY:
Delayed cord clamp of at least 30 seconds in neonates under 37 weeks has shown that these infants have higher circulating blood volume in the first 24 hours, less need for blood transfusions, and less incidence of intraventricular hemorrhage. Delayed umbilical cord clamping has also been shown to increase the initial hematocrit and decrease the need for red blood cell (RBC) transfusions compared with no intervention in infants born between 27 and 33 weeks' gestation. However, a delay in cord clamping of 30-45 seconds may theoretically interfere with neonatal resuscitation. There have been few studies that addressed the active milking of the cord and its effect on neonatal resuscitation. Active milking of the umbilical cord towards the baby prior to clamping (rather than passive) should take less than 5 seconds to perform and should not interfere with neonatal resuscitation. Umbilical cord milking, as an alternative to delayed cord clamping, has been shown to increase the circulatory blood volume expressed as the hemoglobin value. Active milking of the cord prior to clamping, however, is not considered standard of care and only 1 Japanese randomized control study has reported that umbilical cord milking reduces the need for RBC transfusions, thus reducing the number of infants requiring a RBC transfusion as compared with control conditions. Our study aims to test the hypothesis that active milking of the umbilical cord will reduce the need for transfusion in preterm infants.

DETAILED DESCRIPTION:
The proposed design is a randomized controlled trial. Pregnant women at risk for delivering a singleton preterm infant between 24 and 28 weeks gestation will be randomized prior to delivery into one of two treatment arms. Common reasons for needing to be delivered at this early gestational age include but are not limited to: preterm labor not responding to tocolytic medications, incompetent cervix with cervical dilation and no contractions, clinical chorioamnionitis requiring delivery for maternal/fetal benefit, severe preeclampsia, severe growth restriction with a non-reassuring fetal heart rate tracing. The first arm will include active milking of the umbilical cord toward the neonate's umbilicus prior to cord clamping at delivery while the second arm will not include this intervention and will have their respective cord immediately clamped in the usual fashion post delivery (control).

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Delivery anticipated between 24 and 28+6 weeks gestation
* There is enough time from admission to anticipated delivery to properly obtain consent from the patient

Exclusion Criteria:

* Multifetal gestation
* Antenatally diagnosed major congenital anomaly
* Known Rh sensitized pregnancy
* Hydrops fetalis (any etiology)
* Known positive maternal Parvovirus titers
* Elevated peak systolic velocity of the fetal Middle Cerebral Artery (MCA)
* Clinical suspicion of placental abruption at delivery due to excessive maternal bleeding or uterine hypertonicity
* Maternal age under 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Red blood cell transfusion | 28 days
  need for packed red blood cell transfusion in the first 28 days of neonatal life

SECONDARY OUTCOMES:
Volume of blood transfusion | 28 days
  total volume of packed RBC's transfused in first 28 days of neonatal life
Intraventricular Hemorrhage | 28 days
  diagnosis of IVH in first 28 days of neonatal life
Days until transfusion | 28 days
  number of days until first RBC transfusion in first 28 days of life
Respiratory Distress Syndrome | 28 days
  diagnosis of RDS in first 28 days of neonatal life
Retinopathy of Prematurity | 28 days
  diagnosis of ROP in first 28 days of neonatal life
Chronic Lung Disease | 28 days
  diagnosis of CLD in first 28 days of neonatal life
Sepsis | 28 days
  diagnosis of sepsis in first 28 days of neonatal life
Necrotizing Enterocolitis | 28 days
  diagnosis of nec in first 28 days of neonatal life
Apgar scores | 10 minutes
  1, 5, and 10 minute Apgars scores
cord PH | 1 hour
  umbilical cord pH immediately after delivery
Neonatal resuscitation | 1 hour
  Neonatal Resuscitation measures immediately after birth, including intubation, surfactant administration, stimulation, compressions, epinephrine
Initial Hemoglobin/Hematocrit | 1 day
  Initial neonatal H/H
Initial blood pressure | 1 day
  Initial neonatal blood pressure
Neonatal jaundice | 28 days
  Need for bili lights to treat neonatal jaundice, maximum total bilirubin, number of days of bili lights
Neonatal death | 28 days
  Incidence of neonatal death in the first 28 days of life, age of neonate at death
Length of admission | 28 days
  Length of neonatal admission (up to 28 days)
Length of intubation | 28 days
  Length of need for neonatal intubation in first 28 days of life
Periventricular Leukomalacia | 28 days
  diagnosis of PVL in first 28 days of neonatal life
Hyperkalemia | 28 days
  diagnosis of Hyperkalemia in first 28 days of neonatal life

CONTACTS AND LOCATIONS:
Overall Officials: Margarita deVeciana, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States